CLINICAL TRIAL: NCT02605616
Title: A Randomized, Double-Blinded, Placebo-controlled Phase IIa Study to Assess the Efficacy and Safety of a Novel AstraZeneca Compound in Subjects With Non-alcoholic Steatohepatitis (NASH) or Non-alcoholic Fatty Liver Disease (NAFLD)
Brief Title: Use of a Novel Drug in People With Non-alcoholic Steatohepatitis (NASH) or Non-alcoholic Fatty Liver Disease (NAFLD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Astra Zeneca notified Dr. Rita Basu that they will not manufacture new drug due to business reasons and study was stopped.
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Rita Basu, MD, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-000013
Record Dates: First submitted 2015-09-18; First posted 2015-11-16 (Estimated); Results first posted 2022-04-04 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Non-alcoholic Fatty Liver Disease (NAFLD); Non-alcoholic Steatohepatitis (NASH)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — MeRho-Az compound

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active drug AZ compound (Experimental): AZ compound 800 mg/day for 12 weeks (plus or minus 1 week) in two divided doses morning (400 mg) and evening (400 mg).
  Interventions: Drug: AZ compound
- Placebo (Placebo Comparator): Placebo 800 mg/day for 12 weeks (plus or minus 1 week) in two divided doses morning (400 mg) and evening (400 mg).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AZ compound — AZ compound 800 mg/day for 12 weeks (plus or minus 1 week) in two divided doses morning (400 mg) and evening (400 mg).
  Arms: Active drug AZ compound
Other: Placebo — Placebo 800 mg/day for 12 weeks (plus or minus 1 week) in two divided doses morning (400 mg) and evening (400 mg).
  Arms: Placebo

SUMMARY:
Does the novel drug decrease liver fat in subjects with NASH or NAFLD as compared to placebo

DETAILED DESCRIPTION:
We propose to evaluate hepatic fat and hepatic fibrosis using magnetic resonance elastography (MRE) liver (pre vs. post). We will also establish glucose tolerance status by our established labeled oral glucose tolerance test (OGTT) (6,6 ²H2 glucose). Following baseline evaluation subjects with biopsy/MRE proven NASH will be randomized to one of two groups and treated either with active drug (AZ compound) or placebo for 12 weeks (plus or minus 1 week). Subjects with history suggestive of non-alcoholic fatty liver disease (NAFLD) or NASH will be invited to participate. If they meet criteria following initial screening they will be included in the study. OGTT, liver MRE will be repeated. Liver enzymes [aspartate aminotransferase (AST), alanine aminotransferase (ALT),alkaline phosphatase (ALP)] as well as other safety tests [creatine phosphokinase (CPK), thyroid stimulating hormone (TSH), international normalized ratio (INR),total bilirubin] will be measured before, monthly during therapy and at one month following therapy. Furthermore, we will also do the subgroup analysis in NASH/NAFLD subjects with and without diabetes to see the effect of the drug.

ELIGIBILITY:
Inclusion Criteria:

* Age: 21-75
* Body Mass Index (BMI) >19 kg/m^2
* Subjects with biopsy/MRE proven NASH [MRE liver fat ≥ 5%, with elevated liver enzymes ALT <5x upper limit normal (ULN)].
* Subjects with NAFLD and MRE shows F0 or greater fibrosis
* Subjects with history suggestive of NAFLD/NASH
* Total bilirubin must be < 1.5 x ULN and INR must be < 1.3 at baseline screening.
* TSH and CPK will be within normal limits (WNL) at screening.
* Subjects with type 2 diabetes who are on stable doses of medications (except pioglitazone) to control hyperglycemia and have baseline HbA1c of 10% or lower.
* Hemoglobin must be greater than or equal to 12.0 in males and 11.0 in females.

Exclusion Criteria:

* Medications that may affect glucose metabolism such as corticosteroids, opiates, barbiturates, and anticoagulants.
* Subjects with anemia, and symptoms suggestive of undiagnosed illness, overt hepatic disease, stroke, Alzheimer's disease, autoimmune hepatitis, alcoholism or increased alcohol consumption over the American Diabetes Association (ADA) guidelines.
* Any disorder that may potentially impact the outcome measures.
* Pregnant women and children.
* Subjects planning weight loss or in any weight loss program.
* Subjects taking TZD's, Atazanavir, Indinavir, Ketoconazole, Valproic acid, Silybum marianum and Valeriana officinalis.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2015-11; Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rita Basu, MD, Principal Investigator — University of Virginia
Locations (1):
- Yogesh Yadav, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
No: There is not a plan to make IPD available

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Drug AZ Compound | Placebo
Started | 46 | 47
Completed | 42 | 43
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Population: The overall number of baseline participants does not differ from the number assigned to the arm or comparison group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Drug AZ Compound | Placebo | Total
Number analyzed (Participants) | 46 | 47 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (11.7) | 53.3 (11.4) | 53.7 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 29 | 57
  Male | 18 | 18 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 45 | 43 | 88
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 43 | 45 | 88
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 46 | 47 | 93
Number of baseline particpants [Count of Participants; unit: Participants] | 46 | 47 | 93

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Hepatic Fat
Description: Percentage Hepatic fat measured using Magnetic Resonance Imaging (Proton Density Fat Fraction). A cut-off of <5% is used to distinguish between normal and fatty liver.
Time Frame: baseline, approximately 12 weeks
Measure: Mean (Standard Deviation); unit: Percentage change in liver fat fraction
Arm/Group | Active Drug AZ Compound | Placebo
Number analyzed (Participants) | 42 | 43
Percentage change in liver fat fraction | -0.667 (5.246) | 0.139 (4.323)

2. Primary Outcome: Number of Participants With no Conversion of [13C] Cortisone to [13C] Cortisol
Description: Hepatic conversion of [13C] cortisone to [13C] cortisol was assessed before and after the treatment in both groups using the triple tracer cortisol test.
Time Frame: baseline, approximately 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Active Drug AZ Compound | Placebo
Number analyzed (Participants) | 42 | 43
Participants | 42 | 0

3. Secondary Outcome: Liver Fibrosis Measured With MRE in kPa
Description: Liver fibrosis will be measured with Magnetic Resonance Enterography (MRE) at baseline and then compared after ~12 weeks of treatment. A clinical cut-off of 2.93 kPa was used to classify the results as either normal or elevated liver stiffness. Change in Liver fibrosis (kPa) is compared in between the groups.
Time Frame: baseline, approximately 12 weeks
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Active Drug AZ Compound | Placebo
Number analyzed (Participants) | 42 | 43
kPa | -0.639 (0.991) | -0.662 (0.977)

4. Secondary Outcome: Total Insulin Sensitivity (Si) and Hepatic Insulin Sensitivity (Si Liver)
Description: Total insulin sensitivity (Si) and hepatic insulin sensitivity (Si liver) will be measured with an Oral glucose Tolerance test at baseline and after ~12 weeks of treatment.
Time Frame: baseline, approximately 12 weeks
Population: Insulin Sensitivity was measured in the participants that completed the oral glucose tolerance test .
Measure: Mean (Standard Deviation); unit: 10^-4 dl/kg/min per uU/ml
Arm/Group | Active Drug AZ Compound | Placebo
Number analyzed (Participants) | 29 | 32
10^-4 dl/kg/min per uU/ml
  Change in SI | -0.225 (1.918) | 0.719 (3.361)
  Change in Si liver | 0.075 (1.948) | 0.126 (2.369)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Active Drug AZ Compound | Placebo
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/47
Other Adverse Events (participants affected / at risk) | 20/46 | 10/47
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active Drug AZ Compound (N=46) | Placebo (N=47)
Headache (General disorders) | 8 | 4 — Headache
Diarrhea (Gastrointestinal disorders) | 9 | 6
Increased TSH (Endocrine disorders) | 3 | 0

LIMITATIONS AND CAVEATS:
The study was stopped after enrolling 93 patients. The sponsor recalled the batch of AZD4017 /placebo that was provided to the study investigator after the batch of the investigational product failed a routine stability retest that was performed to support potential shelflife extension. Ten patients who were taking either AZD4017 or a placebo were asked to stop taking their drug. Since eight of the10 patients were close to reaching study completion, their data were included in the ITT analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-08): https://cdn.clinicaltrials.gov/large-docs/16/NCT02605616/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/16/NCT02605616/ICF_001.pdf